CLINICAL TRIAL: NCT03797144
Title: A Prospective, Multicenter Evaluation of the CD HORIZON® Fenestrated Screw Spinal System With Fenestrated Screw Cement When Used in the Treatment of Spinal Conditions in Subjects With Compromised Bone Quality
Brief Title: Fenestrated Screw Study
Acronym: FNS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay in enrollment as compared to plan (impacted by COVID-19 pandemic) and availability of data from other data sources to support the products in scope.
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17040SD1703
Record Dates: First submitted 2018-12-14; First posted 2019-01-09 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Degenerative Spinal Disease; Deformity of Spine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fenestrated Screw System (Experimental)
  Interventions: Device: CD HORIZON® Fenestrated Screw System with Fenestrated Screw Cement

INTERVENTIONS:
Device: CD HORIZON® Fenestrated Screw System with Fenestrated Screw Cement — The CD HORIZON® Legacy™ and Solera™ Fenestrated Screw Spinal System consists of a variety of cannulated screws with a series of fenestrations to allow polymethylmethacrylate (PMMA) bone cement (Fenestrated Screw Cement) to be injected into the treated site. The Fenestrated Screw Cement is used to augment screw fixation in subjects with compromised bone quality.

SUMMARY:
The primary objective of this post-market study is to demonstrate that Oswestry disability index (ODI) score improved significantly at 12 months post-operatively as compared to baseline for each indication (degenerative spinal disease and deformity) in subjects with compromised bone quality, who will receive a surgical procedure requiring posterior stabilization and/or immobilization of one or more spinal segments using CD HORIZON® Fenestrated Screw Spinal System with Fenestrated Screw Cement.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet the following inclusion criteria to participate in this trial:

1. One or more of the following diagnostic indications:

   * Degenerative Spinal Disease (e.g. degenerative disc disease, spondylolisthesis and/or spinal stenosis)
   * Deformity (e.g. degenerative deformity)
2. Degenerative Spinal Disease patients only: Patient has been unresponsive to non-operative treatment for at least three months or has progressive symptoms or signs of nerve root/spinal cord compression while undergoing continued non-operative management.
3. Compromised bone quality defined as a hip DXA scan T-score less than or equal to -1.0 or spine quantitative CT (qCT) actual volumetric bone mineral density threshold of ≤ 120 mg/cm3.
4. Requires a procedure with an instrumented, posterior thoracic and/or lumbar spinal stabilization and/or immobilization.
5. Is scheduled to receive a construct using CD Horizon® Spinal System components with at least one Fenestrated Screw cemented with Fenestrated Screw Cement.
6. At least 22 years old or greater at the time of informed consent.
7. Is able to understand and willing to sign the Patient Informed Consent Form.
8. Is willing and able to undergo the study procedure and perform the follow up visits.

Exclusion Criteria:

A subject will be excluded from participating in this trial for any of the following reasons:

1. Has undergone stabilization and/or fusion procedure at the index or adjacent levels.
2. Will undergo vertebroplasty or kyphoplasty procedure during surgery.
3. Has been diagnosed with cauda equina syndrome.
4. Has been previously diagnosed with clinically significant peripheral neuropathy.
5. Has any degree of permanent neurologic deficit due to the presenting spinal disease (e.g. drop foot or gait deficit).
6. Has obesity defined by BMI greater than or equal to 35kg/m2.
7. Has documented allergy to the materials that will be used in the surgical or any imaging procedure (e.g. titanium alloys, cobalt-chromium-molybdenum alloys and PMMA Fenestrated Screw Cement, contrast medium)
8. Has overt or active bacterial infection, local or systemic, and/or potential for bacteremia.
9. Has a non-correctable spontaneous or therapeutic coagulation disorder or history of coagulation disorder associated with bleeding.
10. Has evolutive cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia) nonreactive to medical treatment.
11. Has any disease (e.g., neuromuscular disease, etc.) that would preclude the potential benefit and/or accurate clinical evaluation of the safety of the spinal implant surgery.
12. Is pregnant or planning to become pregnant during the study duration.
13. Is illiterate or considered vulnerable as per the Investigator's assessment (e.g., participants incapable of judgment, or participants under tutelage).
14. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results*.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium
- Tyks Surgical Hospital, Turku, Finland
- Hôpital de la Pitié Salpétrière, Paris, France
- Greece (2):
  - Athens Medical Center, Marousi, Athens
  - Mediterraneo Hospital, Athens
- IRCCS Istituto Clinico Humanitas di Milano, Rozzano, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study aimed at evaluating overall 100 subjects with around 50 subjects (no less than 48 subjects) in each indication subgroup at approximately 10 study sites in Europe. Due to the premature closure of the study, the number of enrolled subjects was 27 (16 belonging to the degenerative spinal disease group and 11 to the deformity group) in 6 sites in Europe.
Groups:
- Degenerative Spinal Disease: Subjects with compromised bone quality requiring stabilization and/or immobilization of the thoracic and/or lumbar spine for Degenerative Spinal Disease indication, defined as back pain of discogenic origin with degeneration of the disc confirmed by history and radiographic studies (e.g. degenerative disc disease, spondylolisthesis and/or spinal stenosis).
- Deformity: Subjects with compromised bone quality requiring stabilization and/or immobilization of the thoracic and/or lumbar spine for deformity indication (e.g. degenerative deformity).
Period: Enrollment
Arm/Group | Degenerative Spinal Disease | Deformity
Started | 16 | 11
Completed | 12 | 10
Not Completed | 4 | 1
Not completed — Protocol Violation | 4 | 1
Period: Surgery
Arm/Group | Degenerative Spinal Disease | Deformity
Started | 12 | 10
Completed | 11 | 10
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: 3 Month
Arm/Group | Degenerative Spinal Disease | Deformity
Started | 11 | 10
Completed | 9 | 10
Not Completed | 2 | 0
Not completed — Early termination cut-off date | 2 | 0
Period: 12 Month
Arm/Group | Degenerative Spinal Disease | Deformity
Started | 9 | 10
Completed | 1 | 1
Not Completed | 8 | 9
Not completed — Early termination cut-off date | 8 | 9
Period: 24 Month
Arm/Group | Degenerative Spinal Disease | Deformity
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Early termination cut-off date | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degenerative Spinal Disease | Deformity | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (10) | 70.9 (6.6) | 70.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Kg] | 60.8 (13.3) | 66.6 (10.8) | 63.5 (12.2)
Height [Mean (Standard Deviation); unit: cm] | 159.3 (7.3) | 158.6 (8.2) | 159.0 (7.6)
Body Max Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.9 (4.1) | 26.4 (3.6) | 25.1 (4.0)
Duration of conservative treatment [Mean (Standard Deviation); unit: months] | 21.6 (49.0) | 20.9 (22.7) | 21.3 (37.8)
Duration of Back Pain Resulting in Planned Surgery [Mean (Standard Deviation); unit: months] | 13.5 (13.6) | 17.5 (17.9) | 15.4 (15.5)
Duration of Leg Pain Resulting in Planned Surgery [Mean (Standard Deviation); unit: months] | 11.0 (11.4) | 9.2 (6.1) | 10.1 (9.1)
Duration of Other Generalized Pain Resulting in Planned Surgery [Mean (Standard Deviation); unit: months] | 0.0 (0.0) | 12.0 (37.9) | 5.7 (26.2)
Patients with previous surgeries [Number; unit: participants] | 4 | 2 | 6
Bone Density Assessment [Mean (Standard Deviation); unit: T-score] — DXA scan of the Hip. A T-score within 1 SD (+1 or -1) of the young adult mean indicates normal bone density.
  A T-score of 1 to 2.5 SD below the young adult mean (-1 to -2.5 SD) indicates low bone mass.
  A T-score of 2.5 SD or more below the young adult mean (more than -2.5 SD) indicates the presence of osteoporosis. Population: For 3 subjects the Bone Density Assessment was missing, and compromised bone quality was confirmed during surgery.
  T-score
    number analyzed (Participants) | 8 | 10 | 18
    (all) | -1.9 (0.8) | -1.9 (0.8) | -1.9 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in ODI (Oswestry Disability Index) at 12 Months Compared to Baseline
Description: Disability associated with thoracic/lumbar spine conditions was assessed using the Oswestry Low Back Pain Disability Questionnaire, which yields the Oswestry Disability Index (ODI), Version 2.1a.This validated instrument is considered one of the principal condition-specific outcome measures used in the management of spinal disorders. ODI is composed by 10 sections.
  Each section can be scored 0 to 5, 5 being the worst case. The score is calculated by summing the different sections and then doubling the total. Maximum score is 100.
  The results are summarized for 21 subjects who were assessed at Baseline and 2 subjects who completed the 12 month follow-up visit. The 24 months follow-up visit did not have data collected and are not reported. The reported ODI was calculated from two timepoints as the value of the baseline point minus the value of the 12 months time point.
Time Frame: Baseline to 12 months
Population: Due to the premature termination of the study, the number of subjects who completed the 12 month follow-up visit was very low (N=2/21, 9.5%).
Measure: Number; unit: score on a scale
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 1 | 1
score on a scale | 46.0 | 17.8

2. Secondary Outcome: Change in ODI From Baseline at 3 Months Visit
Description: Disability associated with thoracic/lumbar spine conditions was assessed using the Oswestry Low Back Pain Disability Questionnaire, which yields the Oswestry Disability Index (ODI), Version 2.1a. [23]. This validated instrument is considered one of the principal condition-specific outcome measures used in the management of spinal disorders.
  ODI is composed by 10 sections. Each section can be scored 0 to 5, 5 being the worst case. The score is calculated by summing the different sections and then doubling the total. Maximum score is 100.
  The results are summarized for 21 subjects who were assessed at Baseline and 19 subjects who completed the 3 months follow-up visit. The 24 months follow-up visit did not have data collected and are not reported. The reported ODI was calculated from two timepoints as the value of the baseline time point minus the value of the 3 months time point.
Time Frame: Baseline, 3 months
Population: The results are summarized for 21 subjects who were assessed at Baseline and 19 subjects who completed the 3 months follow-up visit.
  The 24 months follow-up visit did not have data collected and are not reported. The reported ODI was calculated from two timepoints as the value of the baseline point minus the value of the 3 months time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline | 49.7 (20.0) | 39.6 (13.0)
  3 Month: number analyzed (Participants) | 9 | 10
  3 Month | 20.9 (24.9) | 23.0 (21.7)
  Change from Baseline: number analyzed (Participants) | 9 | 10
  Change from Baseline | 31.5 (28.9) | 16.6 (19.3)
Statistical Analysis 1: Comparison: Degenerative Spinal Disease; To verify that the improvement of ODI from Baseline to 3 Month was significantly greater than 0 for each indication subgroup the following statistical analyses were planned. The null hypothesis was H0: μ_ODI ≤ 0, and the alternative hypothesis was Ha: μ_ODI > 0 where μ_ODI is the mean improvement of ODI score at 3 months from baseline; Test type: Other — A paired t-test for normally distributed data was performed to test whether the mean improvement from baseline was significantly greater than 0. The normality of the data distribution was assessed with the Shapiro-Wilk test; p = 0.06, t-test, 1 sided
Statistical Analysis 2: Comparison: Deformity; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.012, t-test, 1 sided

3. Secondary Outcome: Change in VAS (Visual Analogue Scale) Back and Leg Pain Score at 3 and 12 Months Follow-up Visit From Baseline
Description: Levels of back pain and leg pain were measured using the Visual Analogue Scales (VAS). Subjects were asked to rate the amount of back pain and leg pain they have had in the last week, where 0 is no pain and 10 is the worst pain possible.
  The results are summarized for 21 subjects who were assessed at Baseline, 19 subjects who completed the 3 months follow up visit and 2 subjects who completed the 12month follow-up visit. The reported VAS was calculated from two timepoints as the value of the baseline point minus the value of the 3 months time point and the value of the baseline minus the value of the 12 months time point.
  The 24 months follow-up visit did not have data collected and are not reported.
Time Frame: Baseline, 3, 12 months
Population: The results are summarized for 21 subjects who were assessed at Baseline,19 subjects who completed the 3 months follow-up visit and 2 subjects who completed the 12 months follow-up visit. The reported VAS was calculated from two timepoints as the value of the baseline point minus the value of the 3 months time point and the value of the baseline minus the value of the 12 months time point.
  The 24 months follow-up visit did not have data collected and are not reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 11 | 10
score on a scale
  Back Pain_Baseline | 4.9 (2.9) | 6.8 (2.3)
  Back Pain_3 Months: number analyzed (Participants) | 9 | 10
  Back Pain_3 Months | 2.0 (2.8) | 1.7 (1.8)
  Back Pain_Change from Baseline at 3 Months: number analyzed (Participants) | 9 | 10
  Back Pain_Change from Baseline at 3 Months | 3.3 (2.6) | 5.1 (3.2)
  Back Pain_12 Months: number analyzed (Participants) | 1 | 1
  Back Pain_12 Months | 2.0 (0.0) | 3.0 (0.0)
  Back Pain_Change from Baseline at 12 Months: number analyzed (Participants) | 1 | 1
  Back Pain_Change from Baseline at 12 Months | 3.0 (0.0) | 0.0 (0.0)
  Leg Pain_Baseline | 7.5 (2.2) | 7.1 (2.2)
  Leg Pain_3 Months: number analyzed (Participants) | 9 | 10
  Leg Pain_3 Months | 0.9 (1.3) | 1.3 (1.8)
  Leg Pain_Change from Baseline at 3 Months: number analyzed (Participants) | 9 | 10
  Leg Pain_Change from Baseline at 3 Months | 6.2 (2.7) | 5.8 (2.5)
  Leg Pain_12 Months: number analyzed (Participants) | 1 | 1
  Leg Pain_12 Months | 0.0 (0.0) | 1.0 (0.0)
  Leg Pain_Change form Baseline at 12 Months: number analyzed (Participants) | 1 | 1
  Leg Pain_Change form Baseline at 12 Months | 6.0 (0.0) | 1.0 (0.0)
Statistical Analysis 1: Comparison: Degenerative Spinal Disease; To verify that the improvement of VAS from Baseline to 3 Month was significantly greater than 0 for each indication subgroup the following statistical analyses were planned. The null hypothesis was H0: μ_VAS ≤ 0, and the alternative hypothesis was Ha: μ_VAS > 0 where μ_VAS is the mean improvement of VAS score at 3 months from baseline; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.002, t-test, 1 sided — Back Pain
Statistical Analysis 2: Comparison: Deformity; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.001, t-test, 1 sided — Back Pain
Statistical Analysis 3: Comparison: Degenerative Spinal Disease; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.001, t-test, 1 sided — Leg Pain
Statistical Analysis 4: Comparison: Deformity; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.001, t-test, 1 sided — Leg Pain

4. Secondary Outcome: Change in EQ-5D 5L (European Quality of Life-5 Dimensions) at 3 and 12 Months From Baseline
Description: The EQ-5D 5L (European Quality of Life-5 Dimensions) self-report questionnaire was used to assess health-related quality of life status. The EQ-5D 5L questionnaire includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels, reflecting "no health problems," "slight health problems," "moderate health problems," "severe health problems," and "extreme health problems." The EQ-5D 5L will be used for calculating EQ-5D index score. The EQ-5D VAS was also utilized to document the subject's self-rated overall health state on a 0 to 100 scale (0 = maximal health-related problems, 100 = minimal health-related problems).
  EQ-5D 5L was calculated from two timepoints as the value of the baseline point minus the value of the 3 months follow-up visit and the value of the baseline point minus the value of the 12 months follow-up visit.
  The 24 months follow-up visit did not have data collected and are not reported.
Time Frame: Baseline, 3, 12 months
Population: The results are summarized for 21 subjects who were assessed at Baseline, 19 subjects who completed the 3 months follow-up visit and 2 subjects who completed the 12 months follow-up visit.
  The 24 months follow-up visit did not have data collected and are not reported. The reported EQ-5D 5L was calculated from two timepoints as the value of the baseline point minus the value of the 3 months time point and the value of the baseline minus the value of the 12 months time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 11 | 10
score on a scale
  Index score_Baseline | 0.24 (0.25) | 0.39 (0.19)
  Index score_3 Months: number analyzed (Participants) | 9 | 10
  Index score_3 Months | 0.66 (0.37) | 0.68 (0.34)
  Index score_Change from Baseline at 3 Months: number analyzed (Participants) | 9 | 10
  Index score_Change from Baseline at 3 Months | 0.43 (0.36) | 0.28 (0.33)
  Index score_12 Months: number analyzed (Participants) | 1 | 1
  Index score_12 Months | 0.910 (0.0) | 0.910 (0.0)
  Index score_Change from Baseline at 12 Months: number analyzed (Participants) | 1 | 1
  Index score_Change from Baseline at 12 Months | 0.423 (0.0) | 0.423 (0.0)
  Health State score_Baseline | 64.8 (20.3) | 57.5 (15.9)
  Health State score_3 Months: number analyzed (Participants) | 9 | 10
  Health State score_3 Months | 72.8 (21.7) | 82.2 (16.5)
  Health State score_Change from Baseline: number analyzed (Participants) | 9 | 10
  Health State score_Change from Baseline | 11.9 (35.8) | 24.7 (20.3)
  Health State score_12 Months: number analyzed (Participants) | 1 | 1
  Health State score_12 Months | 90.0 (0.0) | 70.0 (0.0)
  Health State score_Change from Baseline at 12 Months: number analyzed (Participants) | 1 | 1
  Health State score_Change from Baseline at 12 Months | 50.0 (0.0) | 20.0 (0.0)
Statistical Analysis 1: Comparison: Degenerative Spinal Disease; To verify that the improvement of EQ-5D 5L from Baseline to 3 Month was significantly greater than 0 for each indication subgroup the following statistical analyses were planned. The null hypothesis was H0: μ_EQ-5D 5L ≤ 0, and the alternative hypothesis was Ha: μ_EQ-5D 5L > 0 where μ_EQ-5D 5L is the mean improvement of EQ-5D 5L score at 3 months from baseline; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.174, t-test, 1 sided — Health State Score
Statistical Analysis 2: Comparison: Deformity; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.002, t-test, 1 sided — Health State Score
Statistical Analysis 3: Comparison: Degenerative Spinal Disease; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.003, t-test, 1 sided — Index score
Statistical Analysis 4: Comparison: Deformity; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.012, t-test, 1 sided — Index score

5. Secondary Outcome: Rate of Neurological Success at 12-month Visit
Description: Neurological status is based on 4 sections: motor, sensory, reflexes, and straight leg raising, each comprising several elements. Following scales were used to evaluate neurological status: reflexes (0 = Absent or Trace, 1 = Hyper-reflexic, 2 = Normal), sensory function (Light Touch or Pin Prick L1 to S1; 1 = Absent, 2 = Impaired, 3 = Normal), motor function (using 0-5 scores 0-5 whereas 0= Total Paralysis, 1 = Palpable or Visible Contraction, 2 = Active Movement, Gravity Eliminated, 3 = Active Movement, Against Gravity, 4 = Active Movement, Against Some Resistance and 5 = Active Movement, Against Full Resistance (full strength) and straight leg raise (1 = Positive. Patient experiences radiating leg pain below the knee on elevating the leg between 15° and 70° with the knee extended, 2 = Negative. No pain experienced).
  Overall neurological success will be defined as maintenance or improvement in all sections for time period evaluated (each element must remain the same or improve).
Time Frame: Baseline to 12 months.
Population: 21 subjects were assessed at Baseline,19 subjects completed the 3 months follow-up visit and 2 subjects completed the 12 months follow-up visit. Due to the premature termination of the study, the number of subjects who completed the 12 months follow-up visit was very low (N=2/21, 9.5%).
Measure: Number; unit: score on a scale
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 1 | 1
score on a scale
  Motor Functions_Baseline | 5 | 5
  Motor Functions_12 Months | 5 | 5
  Sensory Functions_Baseline | 3 | 3
  Sensory Functions_12 Months | 3 | 3
  Reflexes_Baseline | 2 | 2
  Reflexes_12 Months | 2 | 2
  Straight Leg Raise_Baseline | 2 | 2
  Straight Leg Raise_12 Months | 2 | 2

6. Secondary Outcome: Rate of Intraoperative Cement Extravasation/Leakage. Patients
Description: The rate of intraoperative cement extravasation/leakage as directly assessed by the physician during the surgery or in the post-operative follow-up with imaging procedures.
Time Frame: Surgery to 12 months.
Population: 21 subjects were assessed at surgery,19 subjects completed the 3 month follow-up visit and 2 subjects completed the 12 months follow-up visit.
Measure: Number; unit: participants
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 11 | 10
participants
  Patients with cement extravasation | 3 | 5
  Patients with symptomatic extravasation | 0 | 0

7. Secondary Outcome: Rate of Intraoperative Cement Extravasation/Leakage. Screws
Description: as for outcome 6
Time Frame: Surgery to 12 months.
Population: as for outcome 6
Measure: Number; unit: Screws
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 11 | 10
Screws
  Number of Cemented Fenestrated Screws | 39 | 97
  Fenestrated Screws with cement extravasation | 3 | 8
  Fenestrated screws with symptomatic cement extravasation | 0 | 0

8. Secondary Outcome: Device and/or Procedure Related Adverse Events Through 12 Months.
Description: The adverse events (AEs) were collected from the spinal surgery up to the study cut-off date of 15 JUL 2020. Adverse event relation to the study procedure and to the device was classified by the investigator and by the sponsor as not related, unlikely, possible, probable and causal relationship.
  For the reporting below, AEs classified as having possible, probable and causal relationship are considered as device and/or procedure related. Sponsor assessment is reported if different from the Investigator assessment
  21 subjects were assessed at Baseline,19 subjects completed the 3 month follow-up visit and 2 subjects completed the 12 month follow-up visit.
Time Frame: Surgery to 12 months.
Population: 21 subjects were assessed at surgery,19 subjects completed the 3 months follow-up visit and 2 subjects completed the 12 months follow-up visit. Adverse events up to 12 month follow-up visits are reported in the Outcome Measure Data Table.
Measure: Number; unit: Events
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 11 | 10
Events
  Adverse Event (AE) | 2 | 8
  Serious Adverse Event (SAE) | 1 | 6
  Serious Adverse Device Effect (SADE) | 1 | 5
  Unexpected Serious Adverse Device Effect (USADE) | 0 | 0
  SAEs Related to Procedure | 0 | 5
  SAEs Related to Access System | 0 | 0
  SAEs Related to Cage/Interbody | 0 | 0
  SAEs Related to Anterior Plate | 0 | 0
  SAEs Related to Bone Grafts and Substitutes | 0 | 1
  SAEs Related to Rods | 0 | 1
  SAEs Related to Fenestrated Screw Cement_Investigator assessment | 0 | 0
  SAEs Related to Fenestrated Screw Cement_Sponsor assessment | 0 | 1
  SAEs Related to Fenestrated Screw(s) | 0 | 0
  SAEs Related to other components of the Fixation (stabilization) System | 1 | 0
  SAEs Related to an underlying condition or disease_Investigator assessment | 0 | 2
  SAEs Related to an underlying condition or disease_Sponsor assessment | 1 | 1
  Not Related SAEs_Investigator assessment | 0 | 0
  Not Related SAEs_Sponsor assessment | 0 | 1

9. Secondary Outcome: Rate of Secondary Spinal Surgeries at Index and/or Adjacent Level(s), Resulting From an AE up to 12 Months After Surgery
Description: When a patient requires additional surgery at the index and/or adjacent level(s), it can be an indicator of insufficient outcomes of the initial surgery.
  Secondary spinal surgical procedures resulted from AE(s) could be classified into four categories: revision, removal, reoperation, and other.
  One subject belonging to the Deformity group underwent a reoperation for a foraminal stenosis at index level L5-S1.
Time Frame: Surgery to 12 months.
Population: 21 subjects were assessed at surgery,19 subjects completed the 3 month follow-up visit and 2 subjects completed the 12 month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 11 | 10
Participants | 0 | 1

10. Secondary Outcome: Radiographic Confirmation of Stabilization of the Pedicle Screw Instrumentation at 12-month Visit.
Description: The surgeon or hospital radiologist reviewed radiographs and or CT's to assess for evidence of instability of the pedicle screw instrumentation at 12 months.
  The following were considered as signs of instrumentation instability:
  * Screw pullout
  * Screw loosening
  * Screw toggle
Time Frame: Surgery to 12 months.
Population: 2 subjects completed the 12 month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 1 | 1
Participants
  Stable Construct | 1 | 1
  Unstable Construct | 0 | 0

11. Secondary Outcome: Radiographic Fusion at 12-month Visit for Those Subjects Where Fusion Was Intended.
Description: The surgeon or hospital radiologist determined fusion status for those subjects where fusion was intended. The fusion assessment for each subject was collected at 12 months, preferably by collecting a CT-scan, alternatively fusion could also be collected through X-rays.
  The criterion for fusion when assessed through a CT-scan is bony bridging and when assessed through X-rays the criteria bony bridging, no motion (<4˚) in Flexion/Extension views, and integrity of the instrumentation (implanted devices). A partial fusion (not meeting these criteria) should have been recorded as "No fusion success". For multi-level subjects, fusion success was assessed for each level and overall fusion status was defined as achieving fusion at all treated levels. If one level's fusion status could not be determined, then the subject level was considered unable to determine.
Time Frame: Surgery to 12 months.
Population: 2 subjects who completed the 12 month follow-up visit were analyzed for fusion assessment with radiographic images.
Measure: Count of Participants; unit: Participants
Arm/Group | Degenerative Spinal Disease | Deformity
Number analyzed (Participants) | 1 | 1
Participants
  Fusion success | 0 | 0
  No fusion success | 0 | 0
  Unable to determine | 1 | 1

12. Secondary Outcome: For Deformity Subjects Only: Change in Sagittal Spinopelvic Parameters From Baseline at the 12-month Visit.
Description: Collection of spinopelvic parameters can show if patient's spine is balanced or not prior to and after surgery.
  Any evolution of parameters after the surgery can indicate a change in spinopelvic alignment or a mechanism of regulation/compensation due to an evolution of the spinal alignment.
  The following spinopelvic alignment parameters were assessed in the deformity patients on standing, frontal and sagittal full spine X-ray:
  * Sagittal alignment - Regional parameters: Thoracic Kyphosis (TK), Thoracolumbar kyphosis (TLK), and Lumbar lordosis (LL).
  * Sagittal spinopelvic parameters: Pelvic Incidence (PI): Pelvic Tilt (PT) and Sacral Slope (SS)
Time Frame: Baseline to 12 months
Population: 1 subject who completed the 12 month follow-up visit was analyzed.
Measure: Number; unit: Degrees
Arm/Group | Deformity
Number analyzed (Participants) | 1
Degrees
  Baseline Thoracic Kyphosis (TK) (degrees) | 66
  12-months Thoracic Kyphosis (TK) (degrees) | 78
  Baseline Thoracolumbar kyphosis (TLK) (degrees) | 41
  12-months Thoracolumbar kyphosis (TLK) (degrees) | 5
  Baseline Lumbar lordosis (LL) (degrees) | 50
  12-months Lumbar Lordosis (LL) (degrees) | 58
  Baseline Pelvic Incidence (PI) (degrees) | 46
  12-months Pelvic Incidence (PI) (degrees) | 50
  Baseline Pelvic Tilt (PT) (degrees) | 23
  12-months Pelvic Tilt (PT) (degrees) | 23
  Baseline Sacral Slope (SS) (degrees) | 23
  12-months Sacral Slope (SS) (degrees) | 27

13. Secondary Outcome: For Deformity Subjects Only: Change in Coronal Alignment and Sagittal Vertical Axis From Baseline at the 12-month Visit.
Description: Collection of spinopelvic parameters can show if patient's spine is balanced or not prior to and after surgery.
  Any evolution of parameters after the surgery can indicate a change in spinopelvic alignment or a mechanism of regulation/compensation due to an evolution of the spinal alignment.
  The following spinopelvic alignment parameters were assessed in the deformity patients on standing, frontal and sagittal full spine X-ray:
  * Coronal alignment : Distance between C7 plumb line and the central sacral vertical line
  * Sagittal alignment - Global parameter: Sagittal vertical axis (SVA)
Time Frame: Baseline to 12 months
Population: 1 subject who completed the 12 month follow-up visit was analyzed.
Measure: Number; unit: mm
Arm/Group | Deformity
Number analyzed (Participants) | 1
mm
  Baseline Coronal alignment (mm) | 19.0
  12-months Coronal alignment (mm) | 4.0
  Baseline Sagittal vertical axis (SVA) (mm) | 43.0
  12-months Sagittal vertical axis (SVA) (mm) | 49.0

14. Secondary Outcome: For Deformity Subjects Only: Number of Participants With Coronal Curve Type (T, L, D or N) at Baseline and 12 Months
Description: Collection of spinopelvic parameters can show if patient's spine is balanced or not prior to and after surgery.
  Any evolution of parameters after the surgery can indicate a change in spinopelvic alignment or a mechanism of regulation/compensation due to an evolution of the spinal alignment.
  The following spinopelvic alignment parameter was assessed in the deformity patients on standing frontal full spine X-ray:
  - Coronal Curve Type
  Coronal curve type is determined on the basis of maximal coronal angle measured according to standard Cobb technique and is classified as:
  * Curve type L: patients with a lumbar or thoracolumbar major curve >30˚ (apical level of T10 or lower)
  * Curve type T: patients with a thoracic major curve of >30˚ (apical level of T9 or higher)
  * Curve type D: patients with a double major curve, with each curve >30˚.
  * Curve type N: patients with no coronal curve >30˚.
Time Frame: Baseline to 12 months
Population: 1 subject who completed the 12 month follow-up visit was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Deformity
Number analyzed (Participants) | 1
Participants
  Baseline curve type L | 1
  12-months curve type L | 1
  Baseline curve type T | 0
  12-months curve type T | 0
  Baseline curve type D | 0
  12-months curve type D | 0
  Baseline curve type N | 0
  12-months curve type N | 0

ADVERSE EVENTS:
Time Frame: The adverse events (AEs) were collected from the spinal surgery up to the study cut-off date of 15 JUL 2020 (12 months). At this study cut-off date: - 2 Degenerative Spinal Disease (DSD) patients completed their surgery visit - 8 DSD patients completed up to their 3 month follow-up visit - 1 DSD patient completed up to their 12 month follow-up visit - 9 Deformity patients completed up to their 3-month follow-up visit - 1 Deformity patient completed up to their 12 month follow-up visit
Arm/Group | Degenerative Spinal Disease | Deformity
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 4/10
Other Adverse Events (participants affected / at risk) | 1/11 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degenerative Spinal Disease (N=11) | Deformity (N=10)
SPINAL CSF LEAK (Nervous system disorders) | 0 | 1
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
INCISION WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL FRACTURE AT LEVEL T12 (Injury, poisoning and procedural complications) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degenerative Spinal Disease (N=11) | Deformity (N=10)
PROXIMAL JUNCTIONAL KYPHOSIS (Injury, poisoning and procedural complications) | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
HEMATOMA AT INDEX LEVEL CAUSING FEVER ABOVE 37.8°C (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT03797144/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT03797144/SAP_001.pdf